CLINICAL TRIAL: NCT02376049
Title: An Explorative Clinical Trial to Evaluate an Intra Patient Comparison Design of Topical Agents in Adults With Mild to Moderate Atopic Dermatitis
Brief Title: A Clinical Trial to Compare Topical Agents in Adults With Mild to Moderate Atopic Dermatitis (AD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: EXP-1184
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2017-05

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Eczema; AD
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — pimecrolimus; betamethasone-17,21-dipropionate; Clobetasol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pimecrolimus cream (Active Comparator): Pimecrolimus 1% cream once daily for 14 days
  Interventions: Drug: Pimecrolimus cream
- Betamethasone dipropionate cream (Active Comparator): Betamethasone dipropionate 0.05% cream once daily for 14 days
  Interventions: Drug: Betamethasone dipropionate cream
- Clobetasol propionate cream (Active Comparator): Clobetasol propionate 0.05% cream once daily for 14 days
  Interventions: Drug: Clobetasol propionate cream
- Glaxal Base cream vehicle (Placebo Comparator): Glaxal Base cream vehicle once daily for 14 days
  Interventions: Drug: Glaxal Base cream vehicle

INTERVENTIONS:
Drug: Pimecrolimus cream
  Other Names: Elidel
  Arms: Pimecrolimus cream
Drug: Betamethasone dipropionate cream
  Other Names: Diprosone; Diprolene
  Arms: Betamethasone dipropionate cream
Drug: Clobetasol propionate cream
  Other Names: Dermovate
  Arms: Clobetasol propionate cream
Drug: Glaxal Base cream vehicle
  Other Names: emollient cream
  Arms: Glaxal Base cream vehicle

SUMMARY:
An Explorative Clinical Trial to Evaluate an Intra Patient Comparison Design of Topical Agents in Adults with Mild to Moderate Atopic Dermatitis.

DETAILED DESCRIPTION:
Multi-center, prospective, randomized, vehicle-controlled, investigator-blinded, stable lesion design.

ELIGIBILITY:
Inclusion Criteria:

* Subject with mild to moderate AD
* Four comparable TAs
* TSS of at least 5 on all TAs
* Difference in TSS not greater than 2 between the TAs
* Sign score erythema ≥ 2 between the TAs
* TAs should be at least 2 cm apart

Exclusion Criteria:

* Investigator's opinion
* Fitzpatrick skin type >5
* Topical (i.e. on the TAs) treatment with prohibited medications
* Systemic treatment with prohibited medications
* Phototherapy within prohibited timeframe
* Use of emollients within prohibited timeframe

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Total Sign Score (TSS) change | 14 days
  TSS change at end of treatment in relation to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Emma Guttmann, MD, Principal Investigator — Icahn School of Medicine
Locations (2):
- Innovaderm Research Inc., Montreal, Quebec, Canada
- Beit Harofim, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en